CLINICAL TRIAL: NCT05597852
Title: Feasibility of Integrating Rectal Hydrogel Spacer for Salvage Treatment Using Stereotactic Ablative Body Radiotherapy for Locally Recurrent Prostate Cancer
Brief Title: Using Rectal Hydrogel Spacer for Salvage SABR in Prostate Cancer
Acronym: FIRST STAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: FIRST STAR
Record Dates: First submitted 2022-10-17; First posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients with local recurrence of prostate cancer with previous irradiation will have a hydrogel spacer, SpaceOAR™ inserted.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Arm (Experimental): All patients with local recurrence of prostate cancer post irradiation will undergo placement of a hydrogel spacer between the prostate and rectum, in an effort to decrease toxicity and improve patient's bowel quality of life prior to SABR.
  Interventions: Device: SpaceOAR

INTERVENTIONS:
Device: SpaceOAR — SpaceOAR hydrogel spacer between the prostate and rectum, in an effort to decrease toxicity and improve patient's bowel quality of life.

SUMMARY:
There are several single institutional series that have reported their experience with salvage radiotherapy options that include EBRT, LDR and HDR brachytherapy. Gastrointestinal (GI) toxicity with salvage radiotherapy range between14-58%, respectively for patients undergoing re-irradiation. There is a concern for an increased risk of fistula development in these patients who receive second course of radiation. Hypofractionation using SABR has been utilized in the re-irradiation setting for prostate cancer with good tumor control and toxicity outcomes. In order to decrease the rectal toxicity, dose to the rectum should be kept as low as possible. Several techniques can be used to achieve this: tighter dosimetric dose painting, better patient or organ immobilization or use of a biodegradable gel. The Investigators ropose a phase I study to assess placement of a hydrogel spacer between the prostate and rectum, in an effort to decrease toxicity and improve patient's bowel quality of life.

DETAILED DESCRIPTION:
Primary treatment of prostate cancer includes surgery or radiotherapy. Although significant improvements have been made in patient selection and treatment planning, local recurrence remains a common problem.

In the case of local recurrence after radiation, salvage options may include prostatectomy, salvage external beam radiotherapy (EBRT) or brachytherapy with low-dose (LDR) or high-dose rate (HDR) implantation, cryotherapy and high intensity focused ultrasound.

There are several single institutional series that have reported their experience with salvage radiotherapy options that include EBRT, LDR and HDR brachytherapy (2-7). Rates of grade 2 or higher genitourinary (GU) and gastrointestinal (GI) toxicity with salvage radiotherapy range between 36-50% and 14-58%, respectively for patients undergoing re-irradiation. GI Toxicity, however, is dependent on total rectal dose. This is especially important among patients who are being considered for re-irradiation. There is a concern for an increased risk of fistula development in these patients who receive second course of radiation although with salvage brachytherapy that risk was only 2% and seen only in patients who had a surgical intervention after salvage brachytherapy.

Hypofractionated regimens have become increasingly common in treatment of prostate cancer, especially with advancement of immobilization and imaging techniques that allow smaller margins and daily verification. Hypofractionation using SABR (Stereotatic Ablative Body Therapy) has been utilized in the re-irradiation setting for prostate cancer with good tumor control and toxicity outcomes. In order to decrease the rectal toxicity, dose to the rectum should be kept as low as possible. Several techniques can be used to achieve this: tighter dosimetric objectives, dose painting, better patient or organ immobilization or use of a biodegradable gel. The latter has been used to increase the distance between the prostate and the rectum for patients who are undergoing prostate radiotherapy. Placement of a hydrogel spacer between the prostate and the rectum has been proven in a randomized controlled trial to reduce rectal dose resulting in decreased acute and long-term rectal toxicity and improvement in bowel-related quality of life. SpaceOAR is an FDA and Health Canada approved, commercially available rectal spacer that, when placed between the prostate and the rectum, has demonstrated to greatly reduce rectal dose and toxicity for patients undergoing external beam radiation and LDR brachytherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and radiologically confirmed locally recurrent prostate adenocarcinoma
* Willing to give informed consent to participate in this clinical trial
* Able and willing to complete EPIC and EQ-5D questionnaires

Exclusion Criteria:

* Contraindication to prostate MRI
* Anticoagulation medication (if unsafe to discontinue)
* Diagnosis of bleeding diathesis
* Poor baseline urinary function defined as International Prostate Symptom Score (IPSS) >20
* Evidence of castrate resistance (defined as PSA > 3 ng/ml while testosterone is < 0.7nmol/l). Patients could have been on combined androgen blockade but are excluded if this was started due to PSA progression.
* Definitive extrapelvic nodal or distant metastatic disease on staging investigations.
* Prior ultra-hypofractionated radiotherapy ( SBRT of 5Gy/fraction or higher)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only male patients with Prostate Cancer
Enrollment: 10 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of SpaceOAR | 5 year
  To assess the feasibility, defined as successful placement in 70% of patients, of placing a hydrogel spacer, SpaceOAR™ in patients with biopsy confirmed locally recurrent prostate cancer, undergoing re-irradiation with hypofractionated external beam radiotherapy;

SECONDARY OUTCOMES:
Acute and late cumulative incidence of toxicities | 5 years
  Acute and Late Cumulative incidence Using the CTCAE V5.0 for toxicities. Change of toxicity measured from Baseline
Quality of Life using EPIC | 5 years
  Acute and late quality of life using Expanded Prostate Index Composite (EPIC) Each question is scored from 1-5, 1 being the better outcome and 5 being the worst outcome.
Biochemical disease-free survival | 5 years
  PSA levels will checked for biochemical disease-free survival
Use of salvage ADT | 18 Months
  Up to eighteen months of luteinizing-hormone releasing hormone agonists or antagonists can be used according to physician discretion.
Health utilities | 5 years
  Health utilities using the EuroQol-5D (EQ-5D) Each question is scored from 1-5, 1 being the better outcome and 5 being the worst outcome.
Quality of Life using IPSS | 5 years
  Acute and late quality of life using International Prostate Symptom Score (IPSS) Each question is scored from 1-5, 1 being the better outcome and 5 being the worst outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Amandeep Taggar, MD, Principal Investigator — Sunnybrook
Locations (1):
- Sunnybrook Odette Cancer Centre, Toronto, Ontario, Canada